CLINICAL TRIAL: NCT05222685
Title: Better Together Physician Coaching: An Innovative Solution to Medical Trainee Burnout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 22-0028
Record Dates: First submitted 2022-01-18; First posted 2022-02-03 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Burnout, Professional
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial will offer the intervention group the intervention of BT coaching during the first 6-months while the control group, or "waitlist group" will receive no intervention aside from the usual wellness activities of their institution.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Will receive the 6 month online group coaching program from 9/1/2022-3/1/23
  Interventions: Behavioral: Better Together Physician Coaching
- Control Group (No Intervention): Control group - no coaching intervention from 9/1/2022-3/1/23.
  (They will receive the coaching intervention after study completion from 3/1/23-9/1/23)

INTERVENTIONS:
Behavioral: Better Together Physician Coaching — Professional group coaching for medical trainees. A 6 month, online, group, positive psychology based coaching program for wellness.
  Arms: Intervention Group

SUMMARY:
Burnout refers to feelings of exhaustion, negativism, and reduced personal efficacy resulting from chronic workplace stress. In healthcare, burnout leads to increased medical errors, poorer patient care and negatively affects professional development and retention. Burnout is a growing problem that begins early in medical training. Women and those underrepresented in medicine (URM) experience a disproportionate amount of burnout likely due to the cognitive load required to manage microaggressions, stereotypes, and harmful socially adopted narratives around efficacy. Professional coaching is a metacognition tool with a sustainable positive effect on physician well-being but typically relies on expensive consultants or time-consuming faculty development, often making it infeasible for medical training programs to offer. To overcome this barrier, the investigators created Better Together Physician Coaching (BT) a 6-month coaching program for women residents at the University of Colorado (CU). BT includes regular online group-coaching, written coaching, and weekly self-study modules delivered by physician life coaches (Co-PIs). A pilot randomized controlled trial (RCT) of 101 BT participants demonstrated a statistically significant improvement in burnout, self-compassion, and imposter syndrome in the intervention group. BT will be scaled up to a national level and evaluated with an RCT mirroring our pilot in 10+ graduate medical education (GME) programs for 1000+ participants coordinated and evaluated by our CU team.

To accomplish this goal, the investigators set the following major objectives for this project:

* Prepare to expand the BT program by teaming with a cohort of diverse physician coaches.
* Implement BT in 10+ GME programs to serve 1000+ trainee participants with deliberate inclusion of institutions with diverse GME trainee populations serving geographically rural and/or medically underserved areas.
* Assess our outcomes: primary: reduce burnout as measured by the Maslach Burnout Index (goal: 10% relative improvement), and secondary: self-compassion, imposter syndrome and moral injury. Outcome generalizability and program feasibility at a national level will also be analyzed, as will participant experience to gain a richer understanding of how BT may help trainees, in particular those URM.
* Advance the field of coaching in GME through innovation and dissemination of evidence-based approaches to GME trainee wellbeing.

DETAILED DESCRIPTION:
Background and Significance:

Burnout refers to feelings of exhaustion, negativism, and reduced personal efficacy resulting from chronic workplace stress. In healthcare, burnout leads to increased medical errors, poorer patient care and negatively affects professional development and retention. Burnout is a growing problem that begins early in medical training. Women and those underrepresented in medicine (URM) experience a disproportionate amount of burnout likely due to the cognitive load required to manage microaggressions, stereotypes, and harmful socially adopted narratives around efficacy. Professional coaching is a metacognition tool with a sustainable positive effect on physician well-being but typically relies on expensive consultants or time-consuming faculty development, often making it infeasible for medical training programs to offer. To overcome this barrier, the investigators created Better Together Physician Coaching (BT) a 6-month coaching program for women residents at the University of Colorado (CU). BT includes regular online group-coaching, written coaching, and weekly self-study modules delivered by physician life coaches (Co-PIs). A pilot randomized controlled trial (RCT) of 101 BT participants demonstrated a statistically significant improvement in burnout, self-compassion, and imposter syndrome in the intervention group. This project will scale Better Together up to a national level and evaluated with an RCT mirroring our pilot in 10+ graduate medical education (GME) programs for 1000+ participants coordinated and evaluated by our CU team.

III. Preliminary Studies/Progress Report:

Within the past year, Co-PIs Drs. Adrienne Mann and Tyra Fainstad (AM, TF) created and implemented Better Together Physician Coaching (Better Together, or BT) at the University of Colorado School of Medicine. BT is a coaching program for female identifying GME trainees at CU and its affiliate hospitals (Denver Health, Rocky Mountain Regional VA Medical Center, and The Children's Hospital). Using coaching techniques, BT challenges long-held paradigms fostered by medical training. BT aims primarily to reduce burnout as measured by the MBI with secondary aims to increase self-compassion, reduce imposter syndrome and decrease moral injury among residents who identify as women.

The Co-PIs (AM, TF) are both certified coaches through The Life Coach School™, a training institution for thought-based coaching. This type of coaching focuses on thoughts and beliefs. It combines a cognitive behavioral therapy (CBT) model with mindfulness-based awareness and integrates theories of acceptance and commitment therapy (ACT), nonattachment, and radical questioning from Socratic and Greek philosophies. BT delivers a robust coaching experience via a 6-month web-based, group-coaching model. This novel program allows residents to participate as actively as they are inclined and able, offering flexibility via multiple modalities of coaching: twice weekly group coaching calls, unlimited anonymous written coaching, and weekly self-study modules that are housed on a secure members-only website.

To study the BT program, the Co-PIs received institutional support from the CU Department of Medicine to conduct a pilot randomized controlled trial (RCT), which included support for professional research assistants to both implement and evaluate the program. A convenience sample of 101 female-identifying CU GME trainees from 12 specialties (IM, Family Medicine, Otolaryngology, Pediatrics, OBGYN, General Surgery, Emergency Medicine, Dermatology, Psychiatry, Medicine-Pediatrics, Pathology, and Neurology) was recruited and randomized to receive the 6-month Better Together Program or no-intervention from January-June 2021. The median participant age was 29 years, and all were female-identifying. Of the 101 participants, 33 (32.7%) were PGY-1, 43 (42.6%) were PGY-2, 18 (17.8%) were PGY-3, and 7 (7%) PGY-4 or greater. Nineteen (19%) of participants were in a surgical residency specialty (general surgery, OBGYN, otolaryngology). There were no significant differences in these characteristics between the intervention and control groups at baseline.

All participants completed a pre-survey assessing burnout with the MBI which defines burnout by three subscales (Emotional Exhaustion (EE), Depersonalization (DP), and Personal Accomplishment (PA) as described above). Each item is a 7-point Likert-type question with a frequency response scale ranging from 0 = never to 6 = every day. Higher scores on the EE and DP, and lower scores on the PA subscales indicate greater burnout. Secondary outcomes included Self-compassion with Self-Compassion Scale Short-form (SCSS) where higher scores indicate greater self-compassion,30 the Young Imposter Syndrome Scale (YISS) where a score of more than 5 out of 8 points is diagnostic for Imposter Syndrome31 and the Moral Injury Symptom Scale (MISS) (score 10-100 points) where higher scores equal more moral injury.32

Participants were randomized to the intervention group, (N=50) or control group (N= 51). The intervention group received the 6-month BT coaching program. The control group received the usual wellbeing curriculum provided by their training program, but no BT intervention. Within the BT coaching group, the most frequent topics of coaching included feedback reception, professional appearance, approval-addiction, deficit hiding, balancing motherhood with residency, and low self-confidence. Participants engaged in the live coaching sessions with curiosity, vulnerability, and authenticity, often bringing highly personal and emotional issues to the sessions and supporting each other through encouragement in the Zoom chat function.

From the pilot RCT, the investigators found that at baseline over half of all participants were experiencing moderate or high burnout, consistent with national data. Participants were also experiencing low-moderate self-compassion (mean = 33.6 out of 60; SD=7.17); imposter syndrome (mean = 5.4 out of 8, where score of 5+ is diagnostic for imposter syndrome; SD=2.13); and moderate moral injury (mean =42.02 out of 100; SD=11.08). At the end of 6 months of coaching, a post-survey was offered to both the intervention and control groups. Of the 101 initial survey respondents, 79 responded to the post-survey (78%). A t-test was used to compare the change in subscale score means from baseline to 6 months in the BT coaching versus control groups for the primary and secondary outcomes.

The results on the MBI showed a statistically significant decrease in the emotional exhaustion (EE) dimension of burnout in the intervention group (p=0.03), and the DP and PA components of burnout both trended toward improvement. Self-compassion improved significantly in the intervention group compared to the control group, and imposter syndrome scores improved in the BT coaching group from 5.4 to 4.2 (p=0.01), effectively improving mean scores out of the range for imposter syndrome in this group. Moral injury also trended towards an improvement in the coaching vs control group from baseline to 6 months (40.7 to 35.6 versus 43.7 to 41.7 in intervention vs control, mean difference -3.84, p 0.10), but was not statistically significant.

Based on these promising findings in our pilot RCT, the investigators propose scaling Better Together to a national level to address the unmet need in GME programs to reduce burnout. The investigators are now preparing for a multi-institutional RCT to serve more female identifying trainees with a focus on those who are URM and practicing in medically underserved communities nationwide. The investigators aim to enroll GME programs with geographic and ethnic diversity as well as representative URM trainees to understand the impact of coaching in this vulnerable population.

This randomized controlled trial will mirror our pilot study in which all participants take a pre-survey with outcome measures, then they will be randomized into an intervention or control arm. The intervention group will receive BT during the first 6-months while the control group, or "waitlist group" will receive no intervention aside from the usual wellness activities of their institution. Then all participants will take a post survey. Finally, the control or "waitlist group" will be offered the 6-mont BT program following completion of the study.

The study will begin in September 2022 with approximately 1000 trainees 10+ participating sites. Following the pre-survey, participants will be randomized to the intervention group or the control group. The intervention group will receive the 6-month BT program from 9/2022-2/2023. All participants will complete the post survey in 2/2023. Participants in the intervention group will be offered opportunities to complete qualitative interviews around the program experience after completion of the program. The control group will then be offered the Better Together program from 3/2023 - 9/2023.

Wrap-up:

The final 3 months will focus on preparing our final results for dissemination and finalizing our sustainability plan as the investigators prepare for our future planned funding model.

ELIGIBILITY:
Inclusion Criteria:

* Medical trainees (residents or fellows)
* Identify as female (including trans women, as well as those who identify as gender non-conforming, non-binary, and gender-queer).

Exclusion Criteria:

* Non medical trainees
* Those who do not identify as female (including trans women, as well as those who identify as gender non-conforming, non-binary, and gender-queer).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Medical trainees (residents or fellows) who identify as women, including trans women, as well as those who identify as gender non-conforming, non-binary, and gender queer.
Enrollment: 1017 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Burnout as defined by the Maslach Burnout Inventory (MBI) | pretest will occur prior to the intervention and post test will occur after the 6 month intervention. A post-post test will occur 6 and 12 months after the intervention is done.
  The Maslach burnout inventory (MBI) is a 22-item measurement of worker burnout which assesses emotional exhaustion (EE), depersonalization (DP), and personal fulfillment (PF) domains. Possible scores range from 0-6 on a Likert scale for each item. Scores of EE ≥ 27 points, DP ≥ 10, and PF <33 would indicate a high degree of burnout. Scores of EE≤18 points, DP≤5 points, and PF≥40 points would indicate a low degree of burnout.

SECONDARY OUTCOMES:
Self-Compassion as defined by Neff's Self Compassion Score Short Form (SCS-SF) | pretest will occur prior to the intervention and post test will occur after the 6 month intervention. A post-post test will occur 6 and 12 months after the intervention is done.
  Neff's Self Compassion Score Short Form (SCS-SF) is a 12-item measurement of self compassion. Possible scores range from 0-6 on a Likert scale for each item, where the higher scale scores indicate greater self-compassion. Scores of 1.0- 2.49 are considered to be low, between 2.5-3.5 to be moderate, and 3.51-5.0 to be high.

OTHER OUTCOMES:
Moral Injury as defined by the Moral Injury Symptom Scale for Health Professions (MISS-HP) | pretest will occur prior to the intervention and post test will occur after the 6 month intervention. A post-post test will occur 6 and 12 months after the intervention is done.
  Moral Injury Symptom Scale for Health Professions (MISS-HP) is a 10-item measurement of moral injury. Possible scores range from 0-5 on a Likert scale for each item, where the higher scale scores indicate greater moral injury. Scores >35(on a possible score range of 10 to 100) are considered high for moral injury symptoms causing moderate to extreme problems with family, social, and occupational functioning.
Imposter Syndrome as defined by Young's Imposter Syndrome Symptoms Scale (YISS) | pretest will occur prior to the intervention and post test will occur after the 6 month intervention. A post-post test will occur 6 and 12 months after the intervention is done.
  Young's Imposter Syndrome Symptoms Scale (YISS) is a 8-item measurement of imposter syndrome. Scoring is yes/no where a score of >5/8 is felt to be positive for imposter syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Tyra Fainstad, MD, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
No sharing.

REFERENCES:
- [Result] Villwock JA, Sobin LB, Koester LA, Harris TM. Impostor syndrome and burnout among American medical students: a pilot study. Int J Med Educ. 2016 Oct 31;7:364-369. doi: 10.5116/ijme.5801.eac4. PMID 27802178
- [Result] Pommier E, Neff KD, Toth-Kiraly I. The Development and Validation of the Compassion Scale. Assessment. 2020 Jan;27(1):21-39. doi: 10.1177/1073191119874108. Epub 2019 Sep 13. PMID 31516024
- [Result] Mantri S, Lawson JM, Wang Z, Koenig HG. Identifying Moral Injury in Healthcare Professionals: The Moral Injury Symptom Scale-HP. J Relig Health. 2020 Oct;59(5):2323-2340. doi: 10.1007/s10943-020-01065-w. PMID 32681398
- [Result] Dahlin ME, Runeson B. Burnout and psychiatric morbidity among medical students entering clinical training: a three year prospective questionnaire and interview-based study. BMC Med Educ. 2007 Apr 12;7:6. doi: 10.1186/1472-6920-7-6. PMID 17430583
- [Result] Dyrbye LN, Shanafelt TD, Gill PR, Satele DV, West CP. Effect of a Professional Coaching Intervention on the Well-being and Distress of Physicians: A Pilot Randomized Clinical Trial. JAMA Intern Med. 2019 Oct 1;179(10):1406-1414. doi: 10.1001/jamainternmed.2019.2425. PMID 31380892
- [Result] Palamara K, Chu JT, Chang Y, Yu L, Cosco D, Higgins S, Tulsky A, Mourad R, Singh S, Steinhauser K, Donelan K. Who Benefits Most? A Multisite Study of Coaching and Resident Well-being. J Gen Intern Med. 2022 Feb;37(3):539-547. doi: 10.1007/s11606-021-06903-5. Epub 2021 Jun 7. PMID 34100238
- [Result] Gazelle G, Liebschutz JM, Riess H. Physician burnout: coaching a way out. J Gen Intern Med. 2015 Apr;30(4):508-13. doi: 10.1007/s11606-014-3144-y. Epub 2014 Dec 20. PMID 25527340
- [Result] Abedini NC, Stack SW, Goodman JL, Steinberg KP. "It's Not Just Time Off": A Framework for Understanding Factors Promoting Recovery From Burnout Among Internal Medicine Residents. J Grad Med Educ. 2018 Feb;10(1):26-32. doi: 10.4300/JGME-D-17-00440.1. PMID 29467969
- [Result] Shaikh AA, Shaikh A, Kumar R, Tahir A. Assessment of Burnout and its Factors Among Doctors Using the Abbreviated Maslach Burnout Inventory. Cureus. 2019 Feb 19;11(2):e4101. doi: 10.7759/cureus.4101. PMID 31057995
- [Derived] Mann A, Shah AN, Thibodeau PS, Dyrbye L, Syed A, Woodward MA, Thurmon K, Jones CD, Dunbar KS, Fainstad T. Online Well-Being Group Coaching Program for Women Physician Trainees: A Randomized Clinical Trial. JAMA Netw Open. 2023 Oct 2;6(10):e2335541. doi: 10.1001/jamanetworkopen.2023.35541. PMID 37792378